CLINICAL TRIAL: NCT04229862
Title: Effect of Head Elevation on LMA Supreme Insertion in Patients Undergoing Transurethral Resection of Bladder Tumor: a Randomized Controlled Trial
Brief Title: Effect of Head Elevation on LMA Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-0020
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Laryngeal Masks; Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation with 14 cm high pillow (Experimental): When inserting laryngeal mask airway, head elevation is performed using a 14 cm high pillow.
  Interventions: Procedure: Laryngeal mask airway insertion
- Evaluation with 7 cm high pillow (Active Comparator): When inserting laryngeal mask airway, head elevation is performed using a 7 cm high pillow.
  Interventions: Procedure: Laryngeal mask airway insertion

INTERVENTIONS:
Procedure: Laryngeal mask airway insertion — Laryngeal mask airway insertion in patients who undergoing transurethral bladder tumor resection

SUMMARY:
The purpose of this study is to compare the first attempt success rate of laryngeal mask airway insertion according to the degree of head elevation.

DETAILED DESCRIPTION:
The purpose of this study is to compare the first attempt success rate of laryngeal mask airway insertion between 7 cm head elevation and 14 cm head elevation in patients who undergoing transurethral bladder tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled transurethral bladder tumor resection under general anesthesia
* 20-79 years of age
* American Society of Anesthesiologists physical status ≤3
* Patients who are voluntarily agreed to this clinical study

Exclusion Criteria:

* History of difficult airway
* Expected difficult airway by physical examination
* Unstable teeth or teeth loss
* Obesity (body mass index ≥ 30)
* Recent history of upper respiratory infection
* Patients who are not fasted or who are at risk of aspiration

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | Immediately after mask airway insertion
  The rate of success at the first attempt of laryngeal mask airway insertion

SECONDARY OUTCOMES:
The percentage of glottic opening score | Immediately after mask airway insertion
  The percentage of glottic opening by fiberoptic view
Laryngeal mask airway insertion-related patient satisfaction | At postoperative 6 hours
  A seven-point Likert scale
Second attempt success rate | Immediately after mask airway insertion
  The rate of success at the second attempt of laryngeal mask airway insertion
Third attempt success rate | Immediately after mask airway insertion
  The rate of success at the third attempt of laryngeal mask airway insertion
Oropharyngeal leak pressure | Immediately after mask airway insertion
  Oropharyngeal leak pressure is measured as follows: After setting the expiratory valve to 30 cmH2O at a fixed gas flow rate of 3 L/min, the maximum inflation pressure is measured when a noise of gas leakage is heard in the oropharynx via a stethoscope.
Reposition rate | After mask airway insertion (up to end of surgery)
  The rate of reposition after laryngeal mask airway insertion when ventilation is ineffective or air leaks
Complications associated with laryngeal mask airway insertion | Up to postoperative 3 days
  Complications related with laryngeal mask airway insertion such as cough, vomit, aspiration, regurgitation, bleeding, laryngospasm, and bronchospasm

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohta M. Head elevation beyond sniffing position - An aid to airway management. J Anaesthesiol Clin Pharmacol. 2018 Apr-Jun;34(2):247-248. doi: 10.4103/joacp.JOACP_173_17. No abstract available. PMID 30104838
- [Background] Katsiampoura AD, Killoran PV, Corso RM, Cai C, Hagberg CA, Cattano D. Laryngeal mask placement in a teaching institution: analysis of difficult placements. F1000Res. 2015 Apr 29;4:102. doi: 10.12688/f1000research.6415.1. eCollection 2015. PMID 26401265
- [Background] Horton WA, Fahy L, Charters P. Defining a standard intubating position using "angle finder". Br J Anaesth. 1989 Jan;62(1):6-12. doi: 10.1093/bja/62.1.6. PMID 2917111
- [Background] Takenaka I, Aoyama K, Iwagaki T, Ishimura H, Kadoya T. The sniffing position provides greater occipito-atlanto-axial angulation than simple head extension: a radiological study. Can J Anaesth. 2007 Feb;54(2):129-33. doi: 10.1007/BF03022009. PMID 17272252
- [Background] Jun JH, Baik HJ, Kim JH, Kim YJ, Chang RN. Comparison of the ease of laryngeal mask airway ProSeal insertion and the fiberoptic scoring according to the head position and the presence of a difficult airway. Korean J Anesthesiol. 2011 Apr;60(4):244-9. doi: 10.4097/kjae.2011.60.4.244. Epub 2011 Apr 26. PMID 21602973
- [Derived] Park JY, Yu J, Hong JH, Hwang JH, Kim YK. Head elevation and laryngeal mask airway Supreme insertion: A randomized controlled trial. Acta Anaesthesiol Scand. 2021 Mar;65(3):343-350. doi: 10.1111/aas.13742. Epub 2020 Nov 28. PMID 33174199